CLINICAL TRIAL: NCT05735925
Title: The Role of Host-microbiota Interplay in Hidradenitis Suppurativa Pathogenesis
Acronym: VERIMMUNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Association pour la Recherche Clinique et Immunologique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A02408-35
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hidradenitis Suppurativa (HS) Patients (Experimental): * Skin swab sampling for bacteriological analysis
  * Four skin biopsies:
  a 6-mm and a 4-mm section skin biopsies on a lesional area (inflammatory nodules) a 6-mm and a 4-mm section skin biopsies on a non lesional area
  - blood sample (16 mL)
  Interventions: Diagnostic Test: Skin Swab & Skin Biopsies & Blood Sample
- Healthy Subjects (No Intervention): blood sample (16 mL)

INTERVENTIONS:
Diagnostic Test: Skin Swab & Skin Biopsies & Blood Sample — These intervention will be necessary to phenotype the immune cells that are present in the skin and blood of HS patients
  Arms: Hidradenitis Suppurativa (HS) Patients

SUMMARY:
Hidradenitis Suppurativa (HS) is a chronic disabling inflammatory skin disorder associated with the development of painful and purulent lesions of the folds (armpits, inguinal folds, sub-mammary glands). HS most often develops in adolescence or young adulthood and is characterized by inflammation of the pilo-sebaceous system, of progressive severity (folliculitis, nodule, abscess, fistula). The pathogenesis of HS is still poorly understood: the fact that patients respond to combinations of antibiotics and/or immunosuppressive treatments suggests that the disease could be due to a dysregulated immune response against microbial skin flora. Unconventional lymphocytes (UL), classically considered being at the interface of innate and adaptive immunity, play an important role in immune protection against microbial flora. But UL dysfunction has also been reported in many autoimmune diseases involving various tissues (joints, digestive tract, skin). The uncontrolled and chronic activation of these UL by skin microbiota could therefore play a role in the pathogenesis of HS.

DETAILED DESCRIPTION:
The aim of this exploratory study is to analyze the interplay between microbiota and the innate and adaptative immune response in the pathogenesis of HS. To better understand this host-microbiota interplay, we will assess the number, frequency and functional phenotypes of the different lymphocyte subsets in HS patients, with a special focus regarding the UL. In the same time, we will assess the diversity and nature of skin microbiota of the same patients. Finally, we will explore the relation between the immune response and the skin microbiota in HS, using correlation analysis (Spearman coefficient).

In this study, HS patients will be their own control for leucocyte phenotyping, cytokine analysis and T Cells Receptor (TCR) sequencing (skin biopsies) and for skin microbiota analysis. Paired (age/sex) healthy volunteers will be controls for gut microbiota analysis and for immunophenotyping of circulating leukocytes (Peripheral Blood Mononuclear Cells (PBMC) analysis).

ELIGIBILITY:
Inclusion Criteria:

* Subject able to read, understand and give documented informed consent
* Subject willing and able to comply with the protocol requirements for the duration of the study
* Subject with health insurance coverage according to local regulations
* For woman with childbearing potential, negative pregnancy test at the inclusion visit Specific criteria for HS patients
* Subject diagnosed with HS for at least 6 months
* Subject diagnosed with moderate-to-severe HS defined by HS PGA≥3
* Subject presenting an HS with inflammatory phenotype defined by the presence of folliculitis, nodules and/or abcesses
* Subject suffering from at least 4 flares/year and presenting 5 active inflammatory lesions (nodules and/or abcesses)

Exclusion Criteria:

* Pregnancy or breast-feeding women
* Subject treated by allergen immunotherapy within 4 weeks before inclusion
* Subject treated by Non-Steroidal Anti-Inflammatory Drugs (NSAID), antibiotics or proton-pump inhibitors within 4 weeks before inclusion
* Subject treated by live (attenuated) vaccine within 4 weeks before inclusion
* Subject treated by anti-viral treatment within 4 weeks before inclusion
* Subject treated by anti-diarrhea treatment including, but not limited to Loperamide
* Subject treated by immunosuppressive/immunomodulatory substances including oral corticosteroid or biological agents within 4 weeks before inclusion
* Subject presenting spondylo-arthritis or Inflammatory Bowel Disease (IBD)
* Subject with a Body Mass Index (BMI)<18.5 or BMI>35
* Subject consuming probiotics or using a specific diet (e.g. gluten free, vegetarian, vegan, intermittent fasting)
* Subject with any additional condition that, in the opinion of the investigator, may interfere with the assessment or put the subject at risk
* Linguistic or mentally incapacity to sign the consent form
* Subject protect by the law (adult under guardianship, or hospitalized in a public or private institution for a reason other than study, or incarcerated)
* Subject in an exclusion period from a previous study or who is participating in another clinical trial using a drug Specific criteria for HS patients
* Subject currently experiencing or having a history of other concomitant skin conditions that would interfere with evaluation of HS
* History of allergic reaction to local anesthetic product
* History of wound healing disorders (e.g. hypertrophic scars, keloids)
* History of extensive armpit surgery
* Subject with known active infection to Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV)
* Subject treated for their HS by systemic therapy, investigational or commercial, approved or off label)
* Subject treated for their HS by immunosuppressants or intralesional corticosteroids within 4 weeks before the inclusion
* Subject treated for their HS by topical antibiotics within 4 weeks before the inclusion
* Subject previously treated with monoclonal antibodies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Number of the different leucocytes subsets | Day 0
  Number of the different leucocytes subsets (unconventional and conventional lymphocytes) in the lesional skin versus non lesional skin Number of the different leucocytes subsets (unconventional and conventional lymphocytes) in the blood of HS patients versus healthy volunteers
Frequency of the different leucocytes subsets | Day 0
  Frequency of the different leucocytes subsets (unconventional and conventional lymphocytes) in the lesional skin versus non lesional skin Frequency of the different leucocytes subsets (unconventional and conventional lymphocytes) in the blood of HS patients versus healthy volunteers
Functional phenotype of the different leucocytes subsets | Day 0
  Functional phenotype of the different leucocytes subsets (unconventional and conventional lymphocytes) in the lesional skin versus non lesional skin Functional phenotype of the different leucocytes subsets (unconventional and conventional lymphocytes) in the blood of HS patients versus healthy volunteers

SECONDARY OUTCOMES:
Quantitative RNA | Day 0
  Quantitative RNA expression of selected cytokines' genes in the lesional skin versus non lesional skin
TCR Sequencing | Day 0
  TCR sequencing in the lesional skin versus non-lesional skin
  * TCR sequencing in the blood of HS patients versus healthy volunteers
  * Correlation between lesional skin and blood clones in the same patient will be searched
Bacterial diversity | Day 0
  Bacterial diversity of microbes from skin flora in lesional skin versus non lesional skin
Bacterial abundance | Day 0
  Bacterial abundance of microbes from skin flora in lesional skin versus non lesional skin
Bacterial diversity | Day 14
  Bacterial diversity of microbes from gut flora in HS patients versus healthy volunteers
Bacterial abundance | Day 14
  Bacterial abundance of microbes from gut flora in HS patients versus healthy volunteers
Presence of bacterial DNA translocation | Day 0
  Presence of bacterial DNA translocation in the blood of HS patients
Description of bacterial DNA translocation | Day 0
  Genus, phyla, species, specific bacteria abundance and overall diversity in the blood of HS patients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology-Hôpital Edouard Herriot, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No